CLINICAL TRIAL: NCT01174680
Title: Cardiogoniometry Zur Früherkennung CAD Symptomatik
Brief Title: Cardiogoniometry for Early Diagnosis of Coronary Artery Disease Symptomatik
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CGM@CAD
Record Dates: First submitted 2010-06-07; First posted 2010-08-04 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2010-08

CONDITIONS: Stable Angina Pectoris
Keywords: cardiogoniometry; stable angina pectoris patients
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients with stable angina pectoris (Experimental): stable patients, who have been admitted to one of the participating centres for an elective coronary angiography
  Interventions: Procedure: cardiogoniometry

INTERVENTIONS:
Procedure: cardiogoniometry — In the course of the project a cardiogoniometry will be carried out during the ambulant or residential hospitalization before the coronary angiography.

SUMMARY:
The register study CGM@CAD will examine whether cardiogoniometry can provide additional information concerning the indication for a diagnostic coronary angiography and if so, which additional value it has. Therefore, an additional cardiogoniometry will be carried out in consecutive patients who have been diagnosed with myocardial ischemia by means of established methods (exercise ECG, stress echocardiography, myocardial scintigraphy, or stress-MRT) and for whom an intracardiac catheter examination is regarded as indicated. The results of the different methods - particularly the results of the exercise ECG and the cardiogoniometry - will be checked against the results of the invasive examination as gold standard and the discharge diagnosis with regards to any correlation.

ELIGIBILITY:
Inclusion Criteria:

* Indication for a coronary angiography
* Age > 18 years
* Patients written informed consent

Exclusion Criteria:

* Patients with known CHD (condition after myocardial infarction and/or angio-graphically proven stenosis > 50% and/ or revascularization )
* Patients with acute coronary syndrome
* Patients with pace maker
* Severe valvular heart defect
* 50% extrasystole
* Patients with dysrhythmia, which make a correct interpretation impossible (e.g. VES, bigeminies and other dysrhythmia with a high impact such as atrial extrasystoles)
* Branch block
* Atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
additional value of cardiogoniometry | at hospital admission
  The protocol defines that the medical examination is to be preformed at hospital adimssion and again at discharge. Aim is to examine if cardiogoniometry can provide additional information for the decision to perform a diagnostic coronary angiography and if so, which additional value it has.
additional value of cardiogoniometry | at hospital discharge
  The protocol defines that the medical examination is to be preformed at hospital adimssion and again at discharge. Aim is to examine if cardiogoniometry can provide additional information for the decision to perform a diagnostic coronary angiography and if so, which additional value it has.